CLINICAL TRIAL: NCT01011036
Title: Effects of Gaba-a-Agonists on Pain Mechanisms: An Experimental Study in Healthy Volunteers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Dr. med. Pascal Vuilleumier, Inselspital Bern, Institut für Anästhesiologie und Schmerztherapie
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 152/09; SNF SPUM no.33CM30_124117
Record Dates: First submitted 2009-11-06; First posted 2009-11-11 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Pain
Keywords: healthy study subjects, no disease
MeSH Terms: conditions — Pain | interventions — Clobazam; Clonazepam; Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Other)
  Interventions: Drug: clobazam; Drug: clonazepam; Drug: tolterodine
- 2 (Other)
  Interventions: Drug: clobazam; Drug: clonazepam; Drug: tolterodine
- 3 (Other)
  Interventions: Drug: clobazam; Drug: clonazepam; Drug: tolterodine

INTERVENTIONS:
Drug: clobazam — test substance
Drug: clonazepam — positive control
Drug: tolterodine — active placebo

SUMMARY:
The investigators will use an intradermal capsaicin injection in the forearm to induce a state of localized pain. This localized pain will be measured by different means, and analysed locally and distally by so called quantitative sensory testing. The primary endpoint of measure is the difference in pain perception with and without benzodiazepines/GABA-Agonists around the injection point of capsaicin. The secondary endpoints are to measure pain modulation locally and distally by different quantitative tests as electricity, pressure pain thresholds, and ice water tests.

The investigators' hypothesis is that clobazam induces higher pain thresholds as placebo and less sedation than the control medication clonazepam.

DETAILED DESCRIPTION:
Background

Neuropathic and nociceptive pain are linked to plastic changes of the central nervous system. These lead to lower pain thresholds. An important component of this neuronal plasticity is a diminished inhibition-control of the neurons on the level of the spine, where an alpha-3 subunit of the glycine receptor plays an important role. Modulation of this receptor subunit with specific and non-specific GABA-Agonists produce antinociception. The new fact is, that a subunit specific medication does not induce sedation in animals. The relationship of pain modulation and Gaba-Agonists is not well studied in humans. The benzodiazepine used in pain therapy in humans is clonazepam, which induces a strong sedation, reason why it is not much used in a chronic pain setting. Clobazam is another GABA-Agonist, which is less sedative. To our knowledge its effects on pain modulation has never been studied in humans.

Objective

The aim is an analysis and description of clobazam on the central pain mechanisms. We will use well known quantitative sensory testing methods therefore.

The primary objective is to gather data about potential clinical use of clobazam in pain therapy. The secondary aim would be to do the same tests on new specific alpha-3 agonists, which are being developed by pharmaceutical industry.

Methods

Quantitative sensory testing is being made after eliciting an area of hyperalgesia on the forearm by capsaicin.

The area of hyperalgesia around the injection point will be the primary issue of this study.

The medication given to our patients will be a cross-over, double blind randomized administration of clobazam, clonazepam (positive control) and tolterodine (active placebo). Quantitative sensory testing will be made before and after study medication administration.

The quantitative sensory testing consists of the area of hyperalgesia around capsaicin injection point, pressure pain elicited with an electronic pressure algometer, ice-water testing of the hand, single and multiple electrical skin and muscle stimulation, pressure-cuff algometry and the side effects of the administered medication with psychomotor testing.

Before we start the study protocol each patient will have a blood sample drawn for genetic testing of the different cytochrome subunits (CYP P450 2C19, 3A4).

ELIGIBILITY:
Inclusion Criteria:

* European males
* 18-55 years old
* non smoking status or less than 10 cigarettes per day
* no disease

Exclusion Criteria

* any medication
* any drug abuse
* diseases of any type

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2009-12; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
area of hyperalgesia on the forearm | 11.2010

SECONDARY OUTCOMES:
Diffuse noxious inhibition control | 11.2010
Pressure cuff algometry | 11.2010
pressure pain | 11.2010
electrical stimulation-temporal summation | 11.2010
psychomotor testing | 11.2010
Pharmacokinetic study: plasmatic concentration measured in regular intervals with blood samples, starting at time zero and ending at time plus 24h after drug administration. | 11.2010
Pharmacodynamic study: Measurement of pharmacodynamic behaviour of our 3 tested substances in relation to sedation score. | 11.2010
Pharmacogenetic study: Measurement of subtype cytochrome P450 CYP3A4 and CYP2C19 by metabolites of midazolam and omeprazol. Genotyping of cytochrome P450 CYP3A4 and CYP 2C19. | 11.2010

CONTACTS AND LOCATIONS:
Overall Officials: Michele Curatolo, Professor, Study Director — University of Bern; Pascal H Vuilleumier, Dr med, Principal Investigator — University of Bern
Locations (1):
- Dep of Anesthesiology and Pain Therapy, University Hospital Bern, Bern, Switzerland

REFERENCES:
- [Derived] Vuilleumier PH, Besson M, Desmeules J, Arendt-Nielsen L, Curatolo M. Evaluation of anti-hyperalgesic and analgesic effects of two benzodiazepines in human experimental pain: a randomized placebo-controlled study. PLoS One. 2013;8(3):e43896. doi: 10.1371/journal.pone.0043896. Epub 2013 Mar 15. PMID 23554851